CLINICAL TRIAL: NCT01864070
Title: Phase I Study of TheraSphere and Everolimus Among Patients With Neuroendocrine Tumors and Liver Only or Liver Dominant Disease
Brief Title: Phase 1 TheraSphere + Everolimus With Neuroendocrine Tumors (NETs) + Liver Only or Liver Dominant Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: BTG International Inc. (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1205
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Liver Cancer
Keywords: Liver cancer; Neuroendocrine tumors; NET; Liver dominant disease; TheraSphere; Yttrium-90; Y-90; Everolimus; Afinitor; Zortress; RAD001; Microspheres
MeSH Terms: conditions — Liver Neoplasms; Neuroendocrine Tumors | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TheraSphere + Everolimus (Experimental): Each cycle is 28 days. Target dose of TheraSphere is fixed at 120 Gy to entire tumor bearing portion of liver given at a single session on Cycle 1 Day 15. The dose of everolimus will be escalated in 2 sequential cohorts of 6 TheraSphere-treated patients each. Starting dose of everolimus is 5 mg by mouth daily for cycles 1 and 2. Patients will receive standard dose of Everolimus at 10 mg PO daily starting cycle 3 day 1.
  Once DLT is defined or dose level 2 has been completed, a dose expansion cohort of 10 patients with advanced low to intermediate grade neuroendocrine tumor will be enrolled.
  At least 1 time a week by phone or at the clinic for up to 30 days after last everolimus dose, study staff will follow up. Patient asked about any side effects they may have had.
  Interventions: Other: TheraSphere; Drug: Everolimus; Other: Phone Call

INTERVENTIONS:
Other: TheraSphere — TheraSphere glass microspheres containing Y-90 injected into catheter, and will deliver 120 Gy to entire tumor bearing portion of the liver given at a single session on Cycle 1 Day 15.
Drug: Everolimus — Starting dose: is 5 mg by mouth daily for cycles 1 and 2. Patients will receive standard dose of Everolimus at 10 mg by mouth daily starting cycle 3 day 1.
  Dose Expansion Cohort Starting Dose: Maximum tolerated dose from dose escalation cohort.
  Other Names: Afinitor; Zortress; RAD001
Other: Phone Call — At least 1 time a week by phone or at the clinic for up to 30 days after last everolimus dose, study staff will follow up. Patient asked about any side effects they may have had. The call should last about 10-15 minutes.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of everolimus with TheraSphere that can be given to patients with advanced NETs that have spread to the liver. The safety of everolimus and TheraSphere will also be studied.

Everolimus is designed to block a protein inside the cancer cells, which is also involved in cancer growth.

TheraSphere is a medical device containing a radioactive material called yttrium-90 (Y-90). Tiny glass beads called microspheres are filled with Y-90 and then injected through an artery directly into the liver. This allows a large dose of radiation to be given directly to the tumor, which may lower the risk of side effects from the radiation to other parts of the body and/or to healthy liver tissue. The radiation from TheraSphere stays in the body and begins to lose its effect within 12 days. The glass microspheres will stay in the body from that point on. The radiation will eventually decay (go away). By the time a participant leaves the hospital, the amount of radiation outside of the body will be low enough to not be a threat to others.

DETAILED DESCRIPTION:
Study Groups:

If patient is are found to be eligible to take part in this study, they will be assigned to a dose level of everolimus based on when they joined this study. Up to 3 dose levels of everolimus will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the low dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. If intolerable side effects are seen, the dose may be lowered. This will continue until the highest tolerable dose of everolimus is found. After that, 10 additional participants will be enrolled at the highest tolerable dose that was found.

All participants will receive the same dose level of TheraSphere.

Study Drug Administration:

Each study cycle is 28 days.

On Day 1 of Cycle 1, 2 weeks before the TheraSphere procedure, patient will start taking everolimus.

Patient will take 1-2 tablets of everolimus by mouth 1 time every day. Patient will take the everolimus tablets with a glass of water in the morning at the same time every day. The tablets should be swallowed whole and not chewed or crushed. The tablets may be taken either always with or always without food.

If patient vomits after taking their dose, they should not take another tablet that day. It is very important that patients take the tablets given to them just as the study doctor tells them and that they do not miss any tablets. If patient does forget to take it one day, they should not take any extra doses the next day. Instead, patient should contact their doctor and ask for advice.

On the days of patient's study visits, they should take their dose of everolimus at the clinic, not at home.

TheraSphere Administration:

About 2 weeks before the TheraSphere procedure, patient will have an angiogram. An angiogram is an imaging test that uses contrast dye to help the doctor look at the body's blood vessels. Patient will be given drugs by vein in their arm or hand to help them relax, but patient will stay awake during the procedure. An area in patient's groin will be numbed with anesthetic.

During the procedure, the doctor will insert a catheter into a blood vessel in patient's groin that leads to their liver. Dye will be injected into the catheter, and a series of x-rays will be taken that will allow the doctor to see the blood vessels in patient's liver. At the end of the procedure, the catheter will be removed from patient's groin area. The x-rays taken will be looked at by patient's doctor to plan for their TheraSphere procedure. The angiogram procedure should take about 1½ to 3 hours.

On Day 15 of Cycle 1, patient will receive TheraSphere. Before the procedure, patient will be given drugs by vein in their arm or hand to help them relax, but patient will stay awake during the procedure. An area in patient's groin will be numbed with anesthetic. Patient may ask the study staff for information about how the anesthesia drugs are given and their risks.

The doctor will insert a catheter into a blood vessel in patient's groin that leads to their liver. Based on the planning from patient's angiogram procedure, the doctor will guide the catheter to the target blood vessel. Once the catheter is in the proper blood vessel, the TheraSphere microspheres containing Y-90 will be injected into the catheter to reach the tumor in the liver. After the TheraSphere microspheres are injected, the catheter will be removed from patient's groin. The entire procedure will take about 1½ to 3 hours.

After receiving the TheraSphere microspheres, patient will stay in the recovery area for several hours so that the staff can check patient for possible side effects. If patient has any serious side effects, they may be admitted to the hospital to be checked on and for treatment, if needed.

Study Visits:

Before all visits, patient must fast starting at midnight the night before.

On Day 1 of Cycle 1, if the tests have not been done in the last 5 days:

* Patient will have a physical exam, including measurement of their weight and vital signs.
* Patient will be asked about any symptoms they may have had and any drugs they may be taking.
* Patient's performance status will be recorded.
* Blood (about 4 tablespoons) will be drawn for routine tests and tumor marker testing.
* Urine will be collected for routine tests.
* If patient's doctor thinks it is needed, blood (about 2 teaspoons) will be drawn to check for hepatitis B and/or C.

On Day 14 or 15 of Cycle 1:

* Patient will have a physical exam, including measurement of their weight and vital signs.
* Patient will be asked about any side effects they may have had.
* Patient's performance status will be recorded.
* Blood (about 3 tablespoons) will be drawn for routine tests.

On Day 1 of Cycles 2 and beyond:

* Patient will have a physical exam, including measurement of their weight and vital signs.
* Patient will be asked about any side effects they may have had and any drugs they may be taking.
* Patient's performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.

On Day 1 of Cycles 2 and 3 and every 3-6 weeks after that, blood (about 2 teaspoons) will be drawn to check for hepatitis B and/or C if the doctor thinks it is needed.

On Day 1 of Cycles 2, 4, and every 3 cycles after that, blood (about 2 tablespoons) will be drawn for tumor marker testing and additional routine tests.

On Day 1 of Cycles 4 and beyond, urine will be collected for routine tests.

On Day 1 of Cycle 4 and every 3 cycles after that, patient will have a CT scan, MRI, and/or x-ray to check the status of the disease.

Length of Dosing:

Patient will receive TheraSphere on Day 15 of Cycle 1 and they may continue taking everolimus for up to 12 cycles, as long as the doctor thinks it is in patient's best interest. Patient will no longer be able to take everolimus if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Patient's participation on the study will be over once they have completed the follow-up.

End-of-Dosing Visit:

Within 1 week after patient stops taking the study drug, the following tests and procedures will be performed. Patient must fast starting at midnight the night before this visit.

* Patient will have a physical exam, including measurement of their weight and vital signs.
* Patient will be asked about any side effects they may have had.
* Patient's performance status will be recorded.
* Blood (about 3 tablespoons) will be drawn for routine tests and tumor marker testing. This blood draw will include a pregnancy test if patient can become pregnant.
* Urine will be collected for routine tests.
* Patient will have a CT scan, MRI, and/or x-ray to check the status of the disease.

Follow-up:

At least 1 time a week by phone or at the clinic for up to 30 days after patient's last everolimus dose, the study staff will follow up with patient. Patient will be asked about any side effects they may have had. The call should last about 10-15 minutes.

If patient left the study because of a side effect, they will continue to be contacted by the study staff until the side effect has gone away or become stable.

This is an investigational study. Everolimus is commercially available and FDA approved to treat advanced pancreatic NETs and other types of cancer. The combination of everolimus and TheraSphere in this study is investigational.

TheraSphere is commercially available and FDA approved as a radiation treatment for liver cancer. The use of TheraSphere in this study is investigational.

Up to 22 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
2. Patients must have histologically or cytologically confirmed low or intermediate grade neuroendocrine tumor, for which standard curative measures do not exist. Patients with neuroendocrine tumors associated with multiple endocrine neoplasia type 1 (MEN1 syndrome) will be eligible.
3. Patients must have liver-only or liver-dominant disease.
4. Patient deemed suitable for TheraSphere therapy after review of anatomic imaging by an Interventional Radiologist.
5. No prior biliary enteric anastomosis.
6. Intact portal vein and hepatic artery.
7. Age >/= 18 years of age.
8. World Health Organization (WHO) performance status of 0 or 1.
9. Patients must have normal organ and marrow function as defined below: a) leukocytes >/= 3,000/mcL; b) absolute neutrophil count >/= 1,500/mcL; c) hemoglobin >/= 9 g/dL*; d) platelets >/= 100,000/mcL; e) total bilirubin </= 1.5 X upper limit of normal (ULN); f) AST (SGOT) and ALT (SGPT) </= 1.5 X institutional ULN (5x if liver function test [LFT] elevations due to liver metastases); g) creatinine </= 1.5 X institutional ULN OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal. *Eligibility level for hemoglobin may be reached by transfusion.
10. The patient must have fasting serum glucose </= 1.3 X upper limit of normal.
11. Fasting serum cholesterol </= 300 mg/dL OR </= 7.75 mmol/L AND fasting triglycerides </= 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
12. The effects of TheraSphere and everolimus on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use highly effective contraception from the time of study enrollment continuing for the duration of study therapy and for 8 weeks after the last dose of TheraSphere and/or everolimus. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and for 8 weeks after stopping treatment. Highly effective contraception is defined as either: 1) Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.];
13. Continuation of # 12: 2) Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment; 3) Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female subjects on the study, the vasectomised male partner should be the sole partner for that subject.]; 4) Use of a combination of any two of the following (a+b or a+c or b+c): a. Use of oral, injected, implanted or other hormonal methods of contraception; b. Placement of an intrauterine device (IUD) or intrauterine system (IUS); c. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
14. Continuation of # 13: In case of use of oral contraception, women should have been stable on the oral agent before taking study treatment. Sexually active males must use a condom during intercourse while taking the drug and for 8 weeks after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomised men in order to prevent delivery of the drug via seminal fluid. Female partners of male patients must also be advised to use one of the following contraception methods: Use of (1) oral, injected, implanted or other hormonal methods of contraception, or (2) intrauterine device (IUD) or intrauterine system (IUS), or (3) prior male/female sterilization.
15. Women of childbearing potential must have a serum pregnancy test within 7 days prior starting study treatment.
16. Patients must have at least one measurable site of disease according to RECIST in liver.
17. Patients may have received prior systemic anti-neoplastic therapy. There are no limitations on the number of prior regimens. At least 28 days must have elapsed since last treatment. Prior somatostatin analogs use is allowed. The patients on 3 months of stable dose of concurrent somatostatin analogs will be allowed to continue while on study treatment.
18. Patients must have international normalized ratio (INR) </= 1.5.

Exclusion Criteria:

1. Patients may not be receiving any other treatment-related investigational agents.
2. Uncontrolled intercurrent illness including but not limited to: a) ongoing or active infection requiring parenteral therapy at the time of study registration; b) liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class B or C) Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. Testing required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection; c) symptomatic congestive heart failure resulting in a resting O2 saturation of < 92% on room air; d) unstable angina or pectoris myocardial infarction within 6 months of start of study drug; e) serious uncontrolled cardiac arrhythmia; f) known severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or oxygen saturation that is 88% or less at rest on room air. Pulmonary function test (PFT) is not required at study entry.
3. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.).
4. Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study.
5. Patients who previously received liver directed therapy, with either radiofrequency ablation (RFA), transarterial hepatic embolization (TACE) with or without chemotherapy must have >/= 60 days elapsed since last treatment.
6. A known history of human immunodeficiency virus (HIV) seropositivity.
7. Chronic treatment with systemic steroids or another immunosuppressive agent.
8. Female patients who are pregnant or breast feeding, or of reproductive potential who are not using effective birth control methods.
9. Patients with a known history of allergic reactions and/or hypersensitivity attributed compounds of similar chemical or biologic composition to everolimus or other rapamycins (sirolimus, temsirolimus).
10. Known history of brain or leptomeningeal metastases.
11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.
12. Patients who have had hormonal therapy (other than replacement) within 4 weeks prior to entering the study.
13. Not recovered from adverse events related to previous treatment (excluding alopecia) to active Common Terminology Criteria for Adverse Events (CTCAE) Ver. 4 </= grade 1.
14. With the exception of tumor common to a single genetic cancer syndrome (ie MEN1, MEN2, von Hippel-Lindau [vHL], tuberous sclerosis complex [TSC] etc), patients with evidence of more than one active malignancy are excluded. Active malignancy is defined as the presence of primary, regional nodal, or distant metastatic neoplasm that has not undergone definitive therapy.
15. The patient has poorly controlled diabetes mellitus. Patients with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within 1.3 X institutional upper limit of normal and that they are on a stable dietary or therapeutic regimen for this condition.
16. Patients who have received prior treatment with everolimus or an mTOR inhibitor (sirolimus, temsirolimus, everolimus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) for Combination of TheraSphere and Everolimus | 56 days
  Dose limiting toxicity (DLT) defined as any toxicity occurring during the first 56 days of therapy with definite, possible or probable attribution to TheraSphere and/or Everolimus and meets CTCAE version 4.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Nageshwara V. Dasari, MBBS, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org